CLINICAL TRIAL: NCT04689581
Title: Comparison of Postoperative Efficacy of Ultrasound-guided Bi-level Erector Spine Plane Block and Combined Pectoral I-II Block in Breast Cancer Surgery
Brief Title: Comparison of Bi-level Erector Spine Plane Block and Combined Pectoral I-II Block in Breast Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Sevim Cesur, DR, Kocaeli University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: KOU KAEK 2018/487
Record Dates: First submitted 2020-12-27; First posted 2020-12-30 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-06

CONDITIONS: Postoperative Pain; Analgesia
Keywords: Regional anaesthesia; Erector spinae plane block; PECs blocks; Breast cancer surgery
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bi-level erector spinae plane block (Experimental): Bi-level ultrasound (US)-guided Erector spinae plane block (ESP) with 30 ml 0.25% bupivacaine at the T2 andT4 vertebral level will performe preoperatively to all patients in the ESP group.
  Interventions: Other: Ultrasound guided bi-level erector spinae plane block
- Modified pectoral nerve block (Experimental): Ultrasound (US)-guided modified pectoral nerve block (PECs) with 30 ml 0.25% bupivacaine will performe preoperatively to all patients in the PECs group.
  Interventions: Other: Ultrasound guided modified pectoral nerve block

INTERVENTIONS:
Other: Ultrasound guided bi-level erector spinae plane block — Bi-level ultrasound (US)-guided Erector spinae plane block (ESP) with 30 ml 0.25% bupivacaine at the T2 andT4 vertebral level will performe preoperatively to all patients in the ESP group.
  Arms: Bi-level erector spinae plane block
Other: Ultrasound guided modified pectoral nerve block — Ultrasound (US)-guided modified pectoral nerve block (PECs) with 30 ml 0.25% bupivacaine will performe preoperatively to all patients in the PECs group.
  Arms: Modified pectoral nerve block

SUMMARY:
In this study, we compared ultrasound-guided modified pectoral nerve (PECS) block and bi level erector spinae plane (ESP) block on postoperative analgesic effect in breast surgery.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, written consent was obtained from all patients. Patients who meet eligibility requirements will be randomized in a 1:1 ratio to bi- level erector spinae plane block and modified pectoral block.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists Classification (ASA) I-II patients
* 18-70 aged patients
* patients who scheuled elective breast cancer surgery

Exclusion Criteria:

* American Society of Anesthesiologists Classification (ASA) III-IV patients
* patients with coagulopathy
* patients with infection at the injection site

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-15 (Actual)

PRIMARY OUTCOMES:
Morphin consumption | during postoperative 24 hour
  Patients in both groups will provide with intravenous patient-controlled analgesia device containing morphine for postoperative analgesia.
numerical rating scale (NRS) | during postoperative 24 hour
  A numerical rating scale (NRS) requires the patient to rate their pain on a defined scale. For example, 0-10 where 0 is no pain and 10 is the worst pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Cesur, MD, Principal Investigator — Kocaeli University
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

REFERENCES:
- See also: Efficacy of erector spinae plane block for analgesia in breast surgery: a systematic review and meta-analysis — http://pubmed.ncbi.nlm.nih.gov/32609389/